CLINICAL TRIAL: NCT01173029
Title: Observational Study of the Polymorphisms of the Renin-angiotensin-aldosterone System and Their Relation to Resistant Systemic Arterial Hypertension and Adverse Cardiovascular Events
Brief Title: Renin-angiotensin-aldosterone System Polymorphisms in Resistant Hypertension and Adverse Cardiovascular Events
Acronym: GENHART
Status: Completed | Type: Observational
Sponsor: Universidade Gama Filho (Other)
Collaborators: Instituto Nacional de Cardiologia de Laranjeiras (Other)
Responsible Party: Principal Investigator, Paulo Roberto Benchimol Barbosa, Head Researcher, Universidade Gama Filho
Other Study IDs: 0204/21.07.08
Record Dates: First submitted 2010-07-29; First posted 2010-07-30 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Systemic Arterial Hypertension; Hypertension Resistant to Conventional Therapy; Myocardial Infarction; Stroke
Keywords: Systemic arterial hypertension; Hypertension Resistant to Conventional Therapy; Genetic polymorphisms; Renin-angiotensin-aldosterone system genetic polymorphism; Risk markers; Adverse events; Acute myocardial infarction; Stroke
MeSH Terms: conditions — Hypertension; Hypertension Resistant to Conventional Therapy; Myocardial Infarction; Stroke | interventions — Sodium Chloride Symporter Inhibitors; Mineralocorticoid Receptor Antagonists; Adrenergic beta-Antagonists; Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists; Calcium Channel Blockers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Resistant Arterial Hypertension: Subjects with systemic arterial hypertension in whom arterial pressure control was not achieved (24hr ambulatory pressure monitoring: mean 24hr systolic pressure >/=130 mmHg or mean 24hr diastolic pressure >/=80mmHg) by non-investigation specialized hypertensive unit care, in spite of appropriate drug treatment regimen with three or more anti-hypertensive drugs including a diuretic. Anti-hypertensive drug treatment was non-investigational and was prescribed at discretion of the physician who performed primary evaluation.
  Interventions: Drug: Anti-hypertensive drug treatment
- Pseudo-resistant Arterial Hypertension: Subjects with systemic arterial hypertension in whom arterial pressure control was achieved (24hr ambulatory pressure monitoring: mean 24hr systolic pressure <130 mmHg and mean 24hr diastolic pressure <80mmHg) by non-investigation specialized hypertensive unit care, with appropriate drug treatment regimen with three or more anti-hypertensive drugs including a diuretic. Anti-hypertensive drug treatment was non-investigational and was prescribed at discretion of the physician who performed primary evaluation.
  Interventions: Drug: Anti-hypertensive drug treatment

INTERVENTIONS:
Drug: Anti-hypertensive drug treatment — Anti-hypertensive drug treatment was non-investigational. Drug regimen, including which drug and the number of drugs prescribed, was left at discretion of the physician who carried primary assistance.
  Other Names: Thiazide Diuretics; Aldosterone receptor antagonist; Beta-blockers; ACE inhibitors; Angiotensin receptor blockers; Calcium channel blockers

SUMMARY:
Renin-angiotensin-aldosterone system (RAAS) polymorphisms influence 24h arterial pressure fluctuation. Resistant systemic arterial hypertension (RSAH) has an increased risk of end organ damage and unfavourable prognosis, whereas pseudo-RSAH usually respond favourably to drug therapy.

To prospectively investigate, in subjects with RSAH in a tropical South American city: 1) Adverse cardiovascular events defined as fatal and non-fatal stroke or acute myocardial infarction (AMI); and 2) the association of RAAS polymorphisms and adverse cardiovascular events in this population.

Study population: 212 hypertensives recruited from primary care assistance (time since first diagnosis of hypertension: 16.5±8.1 years) and without appropriate pressure control, between 2001 and 2006, corresponding to 0.48% of all hypertensives under care (18 new cases/year), 57±10 years old, 66% females. Under drug treatment schedule: three or more drugs including a diuretic. Ninety two randomly selected hypertensives basis had renin-angiotensin-aldosterone system genetic profile determined. Genetic assessment was carried out using a polymerase chain reaction assay amplification technique. The following single nucleotide polymorphisms were analyzed: renin (G1051A), angiotensinogen (M235T), angiotensin converting enzyme-ACE (I/D), angiotensin II type 1 receptor (A1166C), aldosterone synthase (C344T) and mineralocorticoid receptor (G3514C).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with uncontrolled systemic arterial hypertension despite use of three anti-hypertensive drugs, including one diuretic

Exclusion Criteria:

* Secondary causes of systemic arterial hypertension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects of both genders in investigation for resistant systemic arterial hypertension at the Hypertension Unit, whose arterial pressure control was not achieved by primary care assistance despite regular use of three anti-hypertensive drugs, including one diuretic. All subjects received standard drug therapy, aiming at achieving outpatients clinics pressure <140/90mmHg and were re-evaluated up to four weeks later, including 24h ambulatory arterial pressure monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2001-06; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paulo R Benchimol-Barbosa, MD, DSc, Principal Investigator — Universidade Gama Filho; Priscilla Campos, Principal Investigator — Universidade Gama Filho; José Barbosa-Filho, MD, DSc, Study Chair — Universidade Gama Filho; Ivan Cordovil, MD, Study Chair — Instituto Nacional de Cardiologia, Rio de Janeiro
Locations (1):
- Instituto Nacional de Cardiologia, Rio de Janeiro, RH, Brazil

REFERENCES:
- [Result] Benchimol Barbosa PR, Silva PC, Cordovil I, Barbosa-Filho J. Renin-angiotensin-aldosterone system polymorphisms in resistant hypertension and adverse cardiovascular events: GENHART-RIO Study. Eur Heart J 2010;31(suppl 1):243-243.
- [Result] Benchimol-Barbosa PR, Silva PC, Cordovil I, Barbosa-Filho J. Renin-angiotensin-aldosterone system polymorphisms in resistant arterial hypertension: a genetic risk score for adverse cardiovascular events - GENHART-RIO study. Eur Heart J (2011) 32 (suppl 1): 103-103.
- [Result] Campos PS, Benchimol-Barbosa PR, Cordovil I, Gomes-Filho JB, Tura BR. Polimorfismos do sistema renina-angiotensina-aldosterona na hipertensão arterial resistente e desfechos cardiovasculares adversos: Estudo GENHART-RIO. Arq Bras Cardiol; 2010. 95(3 supl. 1): 59-59
- [Result] Campos FV, Benchimol-Barbosa PR, Vilela FD, Miranda CS, Gobbi GN, Barbosa-Filho J, Gondar AF, Barros MV, Lima AB, Cordovil I. Evaluation on the risk of target organ damage based on the genetic profile of AGT 235MT, mineralocorticoid receptor GCC5GG4C and ACE I/D in subjects with resistant hypertension. Circulation. 2008; 118:e223-e223.
- [Result] Vilela FD, Benchimol-Barbosa PR, Zeno CC, Lima AB, Barros M, Campos FV, Miranda CS, Gobbi GN, Barbosa-Filho J, Cordovil I. The resistant hypertension genotypes of the population resident in Rio de Janeiro. Circulation. 2008; 118:e356-e357.
- [Result] Benchimol-Barbosa PR, Varanda-Rosario AD, Rollin-Ornelas M, Vilela FD, Miranda CS, Gobbi GN, Barbosa-Filho J, Cordovil I. Aldosterone synthase C344T polymorphisms determine circadian arterial blood pressure variation in resistant systemic arterial hypertension. Circulation. 2008; 118:e398-e398.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was carried out in outpatient clinics at Instituto Nacional de Cardiologia.
Pre-assignment Details: Participants who have been diagnosed as secondary hypertension were excluded from the trial before assignment to resistant and pseudo-resistant groups.
Groups:
- Resistant Arterial Hypertension: Subjects with systemic arterial hypertension in whom arterial pressure control was not achieved (24h ambulatory pressure monitoring: mean 24h systolic pressure >/=130 mmHg and mean 24h diastolic pressure >/=80mmHg) by non-investigation specialized hypertensive unit care, in spite of appropriate drug treatment regimen with three or more anti-hypertensive drugs including a diuretic.
- Pseudo-resistant Arterial Hypertension: Subjects with systemic arterial hypertension in whom arterial pressure control was achieved (24h ambulatory pressure monitoring: mean 24h systolic pressure <130 mmHg and mean 24h diastolic pressure <80mmHg) by non-investigation specialized hypertensive unit care, with appropriate drug treatment regimen with three or more anti-hypertensive drugs including a diuretic.
Period: Overall Study
Arm/Group | Resistant Arterial Hypertension | Pseudo-resistant Arterial Hypertension
Started | 61 | 31
Completed | 61 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects referred from primary care with diagnosis of resistant arterial hypertension. Each one had a clinical visit scheduled in the center within one week of referral. All were taking two AH drugs plus diuretic.
  ABP was measured in seated position, after 5 min of rest. If the highest average of two measures was >140/90mmHg, subject was admitted.
Groups:
- Total: Total of all reporting groups
Arm/Group | Resistant Arterial Hypertension | Pseudo-resistant Arterial Hypertension | Total
Number analyzed (Participants) | 61 | 31 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 20 | 70
  >=65 years | 11 | 11 | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 52.3 (9.6) | 56.8 (9.0) | 54.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 20 | 60
  Male | 21 | 11 | 32
Region of Enrollment [Number; unit: participants]
  Brazil | 61 | 31 | 92
Renin-Angiotensin-Aldosterone System Polymorphism [Number; unit: participants] — Genetic assessment was carried out using polymerase chain reaction assay amplification. The following single nucleotide polymorphisms were analyzed: renin (G1051A), angiotensinogen (M235T), ACE (I/D), angiotensin II type 1 receptor (A1166C), aldosterone synthase (C344T) and mineralocorticoid receptor (G3514C)
  participants
    Renin (G1051A) GG | 22 | 10 | 32
    Renin (G1051A) GA | 24 | 6 | 30
    Renin (G1051A) AA | 15 | 15 | 30
Renin-Angiotensin-Aldosterone System Polymorphism [Number; unit: participants] — Genetic assessment was carried out using polymerase chain reaction assay amplification. The following single nucleotide polymorphisms were analyzed: renin (G1051A), angiotensinogen (M235T), ACE (I/D), angiotensin II type 1 receptor (A1166C), aldosterone synthase (C344T) and mineralocorticoid receptor (G3514C)
  participants
    ACE (I/D) II | 12 | 7 | 19
    ACE (I/D) ID | 29 | 13 | 42
    ACE (I/D) DD | 20 | 11 | 31
Renin-Angiotensin-Aldosterone System Polymorphism [Number; unit: participants] — Genetic assessment carried out using polymerase chain reaction assay amplification. The following single nucleotide polymorphisms were analyzed: renin (G1051A), angiotensinogen (M235T), ACE (I/D), angiotensin II type 1 receptor (A1166C), aldosterone synthase (C344T) and mineralocorticoid receptor (G3514C)
  participants
    Angiotensin II type 1 receptor (A1166C) AA | 36 | 26 | 62
    Angiotensin II type 1 receptor (A1166C) AC | 24 | 5 | 29
    Angiotensin II type 1 receptor (A1166C) CC | 1 | 0 | 1
Renin-Angiotensin-Aldosterone System Polymorphism [Number; unit: participants] — Genetic assessment was carried out using polymerase chain reaction assay amplification. The following single nucleotide polymorphisms were analyzed: renin (G1051A), angiotensinogen (M235T), ACE (I/D), angiotensin II type 1 receptor (A1166C), aldosterone synthase (C344T) and mineralocorticoid receptor (G3514C).
  participants
    aldosterone synthase (C344T) CC | 24 | 9 | 33
    aldosterone synthase (C344T) TC | 30 | 15 | 45
    aldosterone synthase (C344T) TT | 7 | 7 | 14
Renin-Angiotensin-Aldosterone System Polymorphism [Number; unit: participants] — Genetic assessment was carried out using polymerase chain reaction assay amplification. The following single nucleotide polymorphisms were analyzed: renin (G1051A), angiotensinogen (M235T), ACE (I/D), angiotensin II type 1 receptor (A1166C), aldosterone synthase (C344T) and mineralocorticoid receptor (G3514C)
  participants
    Angiotensinogen (M235T) TT | 24 | 6 | 30
    Angiotensinogen (M235T) MT | 25 | 15 | 40
    Angiotensinogen (M235T) MM | 12 | 10 | 22
Anti-hypertensive treatment [Number; unit: participants] — Anti-hypertensive treatment, including regimen, drug and the number of drugs prescribed, was left at discrtion of the physician who carried primary assiatnce.
  participants | 61 | 31 | 92

OUTCOME MEASURES:

1. Primary Outcome: Strokes, Either Fatal or Nonfatal
Description: Evidence of clinically definite stroke (focal neurological deficits persisting for more than 24 hours) confirmed or not by non-investigational computerized tomography.
  Death was considered to be related to the event if occurring up to 30 days after the acute event.
  Assessment twice an year by active and direct contact to patients or relatives and review of medical records.
Time Frame: up to 10 years
Population: Number of participants was based on input demand at outpatient clinics. Those who provided provided consent for genetic testing were included.
  A post-hoc sampling procedure (power calculation) validated sample size.
Measure: Number; unit: participants
Arm/Group | Resistant Arterial Hypertension | Pseudo-resistant Arterial Hypertension
Number analyzed (Participants) | 61 | 31
participants | 24 | 7
Statistical Analysis 1: Comparison: Resistant Arterial Hypertension vs Pseudo-resistant Arterial Hypertension; Long-term intention-to-treat data analysis: Student 't' tests Yates's corrected Chi-squared or Fisher's exact test, when appropriate Relative risk estimation Cox proportional-hazard model Hardy-Weinberg equilibrium; Test type: Non-Inferiority or Equivalence — Study power calculation was post-hoc based on composite end-point achieved. Number of exposed: 62 Non-exposed to exposed ratio: 0.5 Relative risk worth detecting: 2.5 Attack rate among non-exposed: 23% Alpha risk: 0.05 Calculated power: 89.8%; p = 0.19, Chi-squared, Corrected — not adjusted; 1 degree-of-freedom; Risk Ratio (RR) = 1.7, 95% CI 2-sided [0.7 to 4.1]

2. Secondary Outcome: Composite of Acute Myocardial Infarctions and/or Strokes Either Fatal or Nonfatal
Description: Evidence of clinically definite stroke (focal neurological deficits persisting for more than 24 hours) confirmed or not by non-investigational computerized tomography.
  Evidence of clinically definite acute myocardial infarction (prolonged > 20min chest pain, not relieved by sublingual nitrate, ST-T segment deviation on 12-lead surface ECG, elevation of plasma troponin >0.2 ng/dL 6h following chest pain episode).
  Death was considered to be related to the event if occurring up to 30 days after the acute event.
  Assessment twice an year by active and direct contact to patients or relatives and review of medical records.
Time Frame: up to 10 years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Resistant Arterial Hypertension | Pseudo-resistant Arterial Hypertension
Number analyzed (Participants) | 61 | 31
participants | 34 | 9
Statistical Analysis 1: Comparison: Resistant Arterial Hypertension vs Pseudo-resistant Arterial Hypertension; Long-term intention-to-treat data analysis: Student 't' test Yates' corrected Chi-squared or Fisher's exact test Relative risk estimation Cox proportional-hazard model Hardy-Weinberg equilibrium; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.01, Chi-squared, Corrected — not adjusted; 1 degree-of-freedom; Risk Ratio (RR) = 2.6, 95% CI 2-sided [1.01 to 7.3]
Statistical Analysis 2: Comparison: Resistant Arterial Hypertension vs Pseudo-resistant Arterial Hypertension; Cox proportional hazard model for the composite endpoint (stroke + myocardial infarction) was assessed. By taking pseudo-resistant arterial hypertension as baseline reference, the hazard ratio for the composite endpoint was calculated; Test type: Non-Inferiority or Equivalence — Proportional-risk hypothesis was tested using the correlation between Schoenfeld's residuals and time (Schoenfeld's global test). The correlation rho was -0.08, Chi-squared was 0.12, and p was 0.73. Therefore, the hypothesis of proportional risk was accepted, validating the correct application model; p = 0.04, Regression, Cox — The p-value was adjusted for confounders: Framingham risk score, body mass index, ethnic groups; The actuarial function of events per time since the first diagnosis of arterial hypertension was plotted for both groups; Hazard Ratio (HR) = 2.2, 95% CI 2-sided [1.1 to 4.8]

3. Post Hoc Outcome: Polygenic Risk Score
Description: Among all analyzed, four renin-angiotensin-aldosterone polymorphisms had statistical significance relating to composite endpoint.
  They were: Angiotensinogen, renin, angiotensin II type 1 receptor and aldosterone synthase. Each polymorphism was arbitrarily weighted according to respective presentation in both alleles as follows: zero (low risk homozygosis), one (heterozygosis) and two (high risk homozygosis). In a following step, they were summed up for each subject, thus, creating a polygenic risk score.
  The weights of the polymorphisms were, thus, defined:
  1. Angiotensinogen: MM - zero, MT - one, TT - two
  2. Renin: AA - zero, GA - one, GG - two
  3. Angiotensin II type 1 receptor: CC - zero, AC - one, AA - two
  4. Aldosterone synthase: CC - zero, TC - one, TT - two
  The polygenic risk score value ranges from zero (all low risk polymorphisms in homozygosis) to eight (all high risk polymorphisms in homozygosis).
Time Frame: up to 10 years
Population: Subjects in both resistant systemic arterial hypertension and pseudo-resistant systemic arterial hypertension groups had their respective genetic background scored according to present rule.
Measure: Number; unit: composite enpoint events
Groups:
- Polygenic Score: Zero: Sum of the weights for analyzing polymorphisms equal to zero.
- Polygenic Score: One: Sum of the weights for analyzing polymorphisms equal to one.
- Polygenic Score: Two: Sum of the weights for analyzing polymorphisms equal to two.
- Polygenic Score: Three: Sum of the weights for analyzing polymorphisms equal to three.
- Polygenic Score: Four: Sum of the weights for analyzing polymorphisms equal to four.
- Polygenic Score: Five: Sum of the weights for analyzing polymorphisms equal to five.
- Polygenic Score: Six: Sum of the weights for analyzing polymorphisms equal to six.
- Polygenic Score: Seven: Sum of the weights for analyzing polymorphisms equal to seven.
- Polygenic Score: Eight: Sum of the weights for analyzing polymorphisms equal to eight.
Arm/Group | Polygenic Score: Zero | Polygenic Score: One | Polygenic Score: Two | Polygenic Score: Three | Polygenic Score: Four | Polygenic Score: Five | Polygenic Score: Six | Polygenic Score: Seven | Polygenic Score: Eight
Number analyzed (Participants) | 1 | 1 | 7 | 14 | 28 | 21 | 14 | 5 | 2
composite enpoint events | 0 | 0 | 1 | 3 | 17 | 10 | 8 | 3 | 2
Statistical Analysis 1: Comparison: Polygenic Score: Zero vs Polygenic Score: One vs Polygenic Score: Two vs Polygenic Score: Three vs Polygenic Score: Four vs Polygenic Score: Five vs Polygenic Score: Six vs Polygenic Score: Seven vs Polygenic Score: Eight; Receiver operating characteristic curve analysis for the polygenic score as predictor of composite endpoint (stroke + myocardial infarction); Test type: Superiority or Other; p < 0.01, z test — At an optimal value of >3, polygenic risk score yielded 90% sensitivity and 40% specificity for composite endpoint; Area under receiver operating characteristic curve; C-statistic = 0.66, 95% CI 2-sided [0.56 to 0.76] — The optimal cutoff value for polygenic risk score was set to >3
Statistical Analysis 2: Comparison: Polygenic Score: Zero vs Polygenic Score: One vs Polygenic Score: Two vs Polygenic Score: Three vs Polygenic Score: Four vs Polygenic Score: Five vs Polygenic Score: Six vs Polygenic Score: Seven vs Polygenic Score: Eight; Cox proportional hazard model of the polygenic risk score<=3 and > 3 for the composite endpoint (stroke + myocardial infarction). By taking polygenic risk score<=3, the hazard ratio for the composite endpoint was calculated for polygenic risk score>3; Test type: Superiority or Other; p = 0.04, Regression, Cox — The p-value was adjusted for confounders: Framingham risk score, body mass index, ethnic group; The actuarial function of events per time since the first diagnosis of arterial hypertension was plotted for polygenic risk score<=3 and >3; Hazard Ratio (HR) = 2.9, 95% CI 2-sided [1.2 to 9.2]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected every 1 year. Study subjects were actively contacted either by telephone or by visit to their home places.
Arm/Group | Resistant Arterial Hypertension | Pseudo-resistant Arterial Hypertension
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/31
Other Adverse Events (participants affected / at risk) | 0/62 | 0/31

LIMITATIONS AND CAVEATS:
Drugs prescribed were at the discretion of attending physician. The impact of anti-hypertensive drugs on the outcomes was not assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No